CLINICAL TRIAL: NCT00413465
Title: Renal Plasma Flow During Experimental Human Endotoxemia
Brief Title: Study of Renal Blood Flow During Human Endotoxemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RPF.sa.cim.rh.dk
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2006-12

CONDITIONS: Healthy; Type 2 Diabetes; Endotoxemia
Keywords: Renal Plasma Flow; Endotoxemia; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Endotoxemia | interventions — endotoxin, Escherichia coli

INTERVENTIONS:
Drug: Escherichia Coli Endotoxin

SUMMARY:
The purpose of the present protocol is to study whether endotoxemia will affect the renal blood flow in type 2 diabetics and healthy volunteers.

DETAILED DESCRIPTION:
Many septic patients develop acute renal failure and the risk is higher in patients with diabetes. The pathogenetic mechanisms behind the development of acute renal failure in connection with sepsis is not completely understood. One among many possible explanations is a change in renal hemodynamics. However, it is still largely unknown what happens to the renal plasma flow during human sepsis. In this study we give endotoxin injection (0,3 ng/kg) to type 2 diabetics and healthy controls as an experimental model of sepsis. Renal plasma flow and glomerular filtration rate are measured by DTPA-renography 1 day before before and 1,25 and 6,5 hours after injection of endotoxin. Furthermore WBC, plasma-cytokines,VCAM-1/ICAM-1, endothelin-1, Thromboxane B2, angiotensin 2, renin and PAI-1 are measured on an hourly basis up to 8 hours after endotoxin injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Type 2 diabetes

Exclusion Criteria:

* Renal failure
* Heart failure
* Lung disease

Ages: 25 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2006-11; Study Completion 2007-12

PRIMARY OUTCOMES:
Renal plasma flow, Glomerular filtration rate, Plasma cytokine content, Endotoxemia score, Plasma angiotensin II and renin content, Plasma thromboxane B2 content, Plasma PAI-1 content

SECONDARY OUTCOMES:
Mean arterial pressure, Heart rate, Oxygen saturation, Body temperature,

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sofie Andreasen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Intensiv Care Unit, Rigshospitalet,, Copenhagen, Denmark